CLINICAL TRIAL: NCT02521467
Title: Adjunctive Role of Platelets Rich Fibrin in Palatal Wound Healing After Free Gingival Graft Harvesting - Case Series
Brief Title: Adjunctive Role of PRF After Free Gingival Graft Harvesting - Case Series
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Assistant Lecturer Oral Periodontology Department, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Doaa Adel
Record Dates: First submitted 2015-07-28; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Platelets Rich Fibrin, Palatal Donor Tissue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRF (Active Comparator): Platelets Rich Fibrin
  Interventions: Biological: Platelets Rich Fibrin in healing of palatal donor tissue
- palatal stent (Placebo Comparator): Palatal stent
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Platelets Rich Fibrin in healing of palatal donor tissue — Platelets Rich Fibrin (PRF) is a second generation of platelets concentrate full of growth factors as PDGF, IGF, TGF which had a role in hemostasis fasten the healing and decrease the pain.
  Arms: PRF
Other: Placebo — the other group is a control group, had no biologic in the palatal wound, only palatal stent
  Other Names: Palatal stent
  Arms: palatal stent

SUMMARY:
Free gingival grafts are important to increase zone of attached gingiva and root coverage. This case series reveals role of platelet-rich fibrin (PRF) as adjunctive therapy in palatal wound healing. The superior healing observed at the PRF membrane sites supports its use in accelerating soft-tissue healing. PRF membrane as a palatal bandage is an efficacious approach to protect the raw wound area of a palatal donor site to reduce healing time and patient discomfort.

DETAILED DESCRIPTION:
Introduction:

Free gingival grafts are one of the common treatment modalities used to increase the zone of keratinized tissue (KT) around implants or prior to ridge augmentation and root coverage. The palatal donor sites had many complications as pain, discomfort and healing by secondary intention. Platelets Rich Fibrin (PRF) is a second generation of platelets concentrate full of growth factors fasten the healing and decrease the pain.

Materials and methods:

Ten patients requiring augmentation of KT participated in this case series. The palatal donor sites of 7 of these patients were covered with PRF membranes with a new suturing technique without palatal stent, the other 3 had palatal stent. Palatal tissue will examined clinically after 3, 7, 10 and 14 days. Considerably very fast healing with 0 pain score was observed during one week in the group with PRF.

ELIGIBILITY:
Inclusion Criteria:

* Systemic free, Good oral hygiene and insufficient attached gingiva prior to ridge augmentation

Exclusion Criteria:

* High arched palate, medically compromised

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pain Assessment by Visual Analog Scale (VAS) | 1 week postoperative
  VAS ranged from 0 (no pain ) to 10 (severe pain)
Clinical healing of the palate | 2 weeks postoperative
  color match, consistency and thickness of palate (Composite measure)